CLINICAL TRIAL: NCT00507169
Title: SVT-40776 in Patients Suffering From Overactive Bladder Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Salvat (Industry)
Responsible Party: Medical Director, Laboratorios SALVAT
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 40776ORII/05IA01
Record Dates: First submitted 2007-07-25; First posted 2007-07-26 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Overactive Bladder (OAB)
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — SVT-40776

INTERVENTIONS:
Drug: SVT-40776

SUMMARY:
The study will examine which dose of SVT-40776 is best in terms of efficacy, safety and tolerability compared to placebo and tolterodine

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from OAB for at least 6 months prior to inclusion

Exclusion Criteria:

* Pregnant and breastfeeding women
* Any medical condition or need for co-medication which interferes with the drug under investigation (SVT-40776) or the comparator (tolterodine)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)